CLINICAL TRIAL: NCT05028387
Title: Safety and Acceptability of a Telemedicine Medical Abortion Service Using the "No-test" Protocol In Ukraine and Uzbekistan.
Brief Title: Telemedicine Medical Abortion Service Using the "No-test" Protocol in Ukraine and Uzbekistan.
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: Charitable Foundation Women Health and Family Planning, Ukraine (Unknown); Women's Wellness Center, Uzbekistan (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1053
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2022-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: medical abortion — medical abortion

SUMMARY:
The goal of this study is to pilot and evaluate a telemedicine medical abortion service delivery that allows remote communication between the woman and provider and limits medically unnecessary in-person visits to health or diagnostic centers.

DETAILED DESCRIPTION:
The goal of this study is to pilot and evaluate a telemedicine medical abortion (TMA) service delivery that allows remote communication between the woman and provider and limits medically unnecessary in-person visits to health or diagnostic centers. Providers will provide counseling by phone or video about pregnancy options and give detailed information about the medical abortion process, expected side effects, and where to seek additional care. The provider will then evaluate the woman's eligibility for TMA service by following the no-test protocol and discuss at-home follow-up using a symptom checklist and a high-sensitivity urine pregnancy test. If pre-treatment tests are needed, women will be referred to a nearby diagnostic center and test results will be forwarded to the study provider. Participants will receive medications by mail or courier service or pick them up at the pharmacy or study clinics, take medications as instructed, and complete at-home follow-ups as discussed with the provider.

ELIGIBILITY:
Inclusion Criteria:

* Is pregnant as determined by a pregnancy test or ultrasound (if obtained prior to contacting the study site)
* Has no contraindications to medical abortion
* Has access to a phone
* Is able to take mifepristone on or before 63 days gestation

Exclusion Criteria:

* Medically ineligible for medical abortion
* Gestational age above 63 days based on LMP

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People seeking abortion
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse events resulting from remote provision of medical abortion | 6 weeks
  Adverse events such as regimen non-compliance or medically unnecessary interventions associated with remote provision of medical abortion.

SECONDARY OUTCOMES:
Satisfaction with remote provision of medical abortion | 6 weeks
  Satisfaction with remote provision of medical abortion measures by 5-point Likert scale. We will be using 1-5 score,
  1. very satisfied,
  2. satisfied
  3. neutral
  4. unsatisfied
  5. very unsatisfied,
  Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (4):
- Ukraine (2):
  - Clinic Vrachebnyye Traditsii, Kiev
  - Regional Clinical Hospital of Rehabilitation and Diagnostics of Poltava Regional Council, Poltava
- Uzbekistan (2):
  - Premium Medical Center, Bukhara Medical Institute, Bukhara
  - Tashkent Medical Academy Clinic, Tashkent

IPD SHARING:
Plan to Share IPD: No